CLINICAL TRIAL: NCT01043874
Title: A Phase IV Study of Nilotinib in Patients With Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP) Who Have Suboptimal Molecular Response on Imatinib
Brief Title: Study to Evaluate Nilotinib in Chronic Myelogenous Leukemia (CML) Patients With SubOptimal Response
Acronym: MACS0911
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107FJP01
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-03

CONDITIONS: Philadelphia Chromosome Positive; Chronic Myelogenous Leukemia in Chronic Phase
Keywords: Chronic phase; Chronic myelogenous leukemia; CML; Philadelphia chromosome positive; Ph+; Nilotinib; CML-CP; Suboptimal molecular response
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nilotinib (Experimental): 400 mg BID
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — 400 mg BID
  Other Names: AMN107

SUMMARY:
To evaluate the major molecular response (MMR) rate at 12 months of nilotinib treatment on study in patients with Philadelphia Chromosome Positive (Ph+) chronic myelogenous leukemia in chronic phase (CML-CP) who have a suboptimal molecular response to imatinib at 18 months or later.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age.
2. ECOG 0, 1, or 2.
3. Have been diagnosed with Ph+ CML-CP and receiving imatinib therapy.
4. Patients with suboptimal molecular response to imatinib treatment continued for at least 18 months (first line therapy)

   Suboptimal molecular response defined as all of the following conditions:
   1. Patients who have achieved CCyR (0% Ph+ chromosomes).
   2. Patients who don't achieve MMR (MMR defined as BCR-ABL/ABL ratio of ≤ 0.1% on the International Scale as detected by RQ-PCR).

   The treatment with imatinib defined as:

   Dose of 300 mg or higher daily must be maintained for a minimum of 3 months prior to study entry.
5. Patients who meet the following laboratory tests criteria:

   1. total bilirubin < 1.5 x ULN,
   2. SGOT and SGPT < 2.5 x ULN,
   3. creatinine < 1.5 x ULN,
   4. Serum amylase and lipase ≤ 1.5 x ULN,
   5. Alkaline phosphatase ≤ 2.5 x ULN unless considered tumor related.
   6. Serum potassium, phosphorus, magnesium and calcium ≥ LLN or correctable with supplements prior to the first dose of study drug.
6. Written informed consent prior to any study related screening procedures being performed.

Exclusion Criteria:

1. Prior accelerated phase or blast crisis CML.
2. Previously documented T315I mutations.
3. Presence of chromosomal abnormalities other than Ph+.
4. Previous treatment with any other tyrosine kinase inhibitor except imatinib.
5. Impaired cardiac function including any one of the following:

   1. Complete left bundle branch block
   2. Congenital long QT syndrome or family history of long QT syndrome
   3. History of or presence of significant ventricular or atrial tachyarrhythmias
   4. Clinically significant resting brachycardia (<50 bpm)
   5. QTcF > 450 msec on screening ECG
   6. Use of a ventricular-paced pacemaker
   7. Myocardial infarction during the last 12 months
   8. Other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension, unstable angina).
6. Treatment with strong CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, St John's Wort), and the treatment cannot be discontinued or switched to a different medication prior to starting study drug. See Section 6.4.3 for complete list of these medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-12; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma K.K., Study Director — Novartis Pharma K.K.
Locations (17):
- Japan (17):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Aomori, Aomori
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Gifu, Gifu
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Sayama, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Saga, Saga-ken
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo

REFERENCES:
- [Derived] Miyamura K, Miyamoto T, Tanimoto M, Yamamoto K, Kimura S, Kawaguchi T, Matsumura I, Hata T, Tsurumi H, Saito S, Hino M, Tadokoro S, Meguro K, Hyodo H, Yamamoto M, Kubo K, Tsukada J, Kondo M, Aoki M, Okada H, Yanada M, Ohyashiki K, Taniwaki M. Switching to nilotinib in patients with chronic myeloid leukemia in chronic phase with molecular suboptimal response to frontline imatinib: SENSOR final results and BIM polymorphism substudy. Leuk Res. 2016 Dec;51:11-18. doi: 10.1016/j.leukres.2016.09.009. Epub 2016 Sep 5. PMID 27771544

RESULTS

PARTICIPANT FLOW:
Groups:
- Nilotinib: Nilotinib 400 mg BID
Period: Overall Study
Arm/Group | Nilotinib
Started | 45
Completed | 39
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1
Not completed — Administrative Problems | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nilotinib
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (14.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: MMR Rate at 12 Mos. of Nilotinib Treatment on Study in Patients With Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP) Who Have a Suboptimal Molecular Response to Imatinib at 18 Months or Later.
Description: MMR is defined as BCR-ABL ratio (%) on IS ≤ 0.1% (corresponds to ≥ 3 log reduction of BCR-ABL transcripts from standardized baseline value
Time Frame: 12 months after treatment
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: % participants achieving MMR
Arm/Group | Nilotinib
Number analyzed (Participants) | 45
% participants achieving MMR | 51.1 [35.8 to 66.3]

2. Secondary Outcome: MMR Rate at 24 Months of Nilotinib Treatment on Study in Patients With Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP)
Description: as for outcome 1
Time Frame: 24 months after treatment
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: % participants achieving MMR
Arm/Group | Nilotinib
Number analyzed (Participants) | 45
% participants achieving MMR | 66.7 [51.0 to 80.0]

3. Secondary Outcome: Time to First MMR of Nilotinib in Patients With Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP) .
Description: as for outcome 1
Time Frame: month 24
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Nilotinib
Number analyzed (Participants) | 45
months | 5.19 (5.494)

4. Secondary Outcome: Duration of MMR of Nilotinib in Patients With Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP) .
Description: as for outcome 1
Time Frame: month 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: % participants w/ durable MMR at 24 mos
Arm/Group | Nilotinib
Number analyzed (Participants) | 45
% participants w/ durable MMR at 24 mos | 51.1 [35.8 to 66.3]

ADVERSE EVENTS:
Arm/Group | Nilotinib
Serious Adverse Events (participants affected / at risk) | 7/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=45)
Anaemia (Blood and lymphatic system disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Chronic myeloid leukaemia transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=45)
Anaemia (Blood and lymphatic system disorders) | 4
Eosinophilia (Blood and lymphatic system disorders) | 4
Conjunctivitis (Eye disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 5
Haemorrhoids (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 6
Face oedema (General disorders) | 3
Fatigue (General disorders) | 4
Oedema (General disorders) | 3
Pyrexia (General disorders) | 5
Hepatic function abnormal (Hepatobiliary disorders) | 5
Hyperbilirubinaemia (Hepatobiliary disorders) | 24
Gastroenteritis (Infections and infestations) | 3
Influenza (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 21
Periodontitis (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 14
Amylase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 8
Blood bilirubin increased (Investigations) | 7
Gamma-glutamyltransferase increased (Investigations) | 4
Lipase increased (Investigations) | 11
Decreased appetite (Metabolism and nutrition disorders) | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 17
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 5
Eczema (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial